CLINICAL TRIAL: NCT00306540
Title: A Multicentre, Parallel Group, Randomised, Double Blind, Placebo Controlled Study of the Use of Quetiapine as an Add on Therapy in the Treatment of Post Traumatic Stress Disorder
Brief Title: Use of Quetiapine as an Add on Therapy in the Treatment of Post Traumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU-SEA-0006; D1449L00005
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Placebo Seroquel + existing therapy
  Interventions: Drug: quetiapine fumarate placebo
- 2 (Experimental): Seroquel + existing therapy
  Interventions: Drug: Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate — oral flexible dose
  Other Names: Seroquel
  Arms: 2
Drug: quetiapine fumarate placebo — oral 0 mg
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate how effective quetiapine versus placebo is when added to an existing therapy, in reducing the symptoms of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised and non-hospitalised patients / Veteran or Civilian / Have had symptoms of PTSD for a minimum of 12 months prior to giving consent to the study

Exclusion Criteria:

* History of psychotic condition / quetiapine or other anti-psychotics not worked previously / Taking prohibited medications (mood stabilizers / substance abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinical Administered PTSD Scale (CAPS2)

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAM-D)
Hamilton Anxiety Scale (HAM-A)
Posttraumatic Stress Disorder Checklist (PCL)
Clinical Global Impressions (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Australia Medical Director, MD, Study Director — AstraZeneca
Locations (3):
- Australia (3):
  - Research Site, Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Melbourne, Victoria